CLINICAL TRIAL: NCT07270419
Title: Aneurysmal Subarachnoid Hemorrhage Multi-Omics Research Program (aSAH-Omics) ：A Multicenter Clinical and Mechanistic Study
Brief Title: Aneurysmal Subarachnoid Hemorrhage Multi-Omics Research Program
Acronym: aSAH-Omics
Status: Recruiting | Type: Observational
Sponsor: Xiaolin Chen, MD (Other)
Collaborators: Peking Union Medical College (Other)
Responsible Party: Sponsor-Investigator, Xiaolin Chen, MD, Prof., Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: KY2025-175-01; 2024ZD0539700 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Multi-Omics; Prognosis; Complications; Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) is a life-threatening cerebrovascular emergency with high mortality and disability rates. Despite advances in neuroimaging and interventional techniques, outcomes remain poor for many patients due to complex post-rupture complications such as delayed cerebral ischemia (DCI), pneumonia, and other systemic injuries. These secondary events critically affect neurological recovery, yet their molecular mechanisms are not fully understood.

This multicenter study aims to investigate the biological basis of post-rupture complications and prognosis in patients with aSAH through integrated multi-omics and clinical data analysis. Biospecimens including blood, cerebrospinal fluid, urine, and other relevant tissues will be collected for genomic, transcriptomic, proteomic, metabolomic, and imaging-omic profiling. By linking molecular data with clinical and imaging indicators, the study seeks to identify key pathways and biomarkers associated with secondary injury and outcome heterogeneity.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (aSAH) is a severe cerebrovascular emergency caused by the rupture of an intracranial aneurysm. Despite advances in neuroimaging and microsurgical or endovascular techniques, aSAH remains associated with high mortality and long-term disability. Post-rupture complications-such as delayed cerebral ischemia (DCI), pneumonia, and other systemic complications-are major determinants of neurological recovery and prognosis.

Following aneurysm rupture, a cascade of complex secondary injuries is triggered, critically influencing clinical outcomes. Beyond the initial hemorrhagic insult, secondary pathophysiological processes-including neuroinflammation, endothelial dysfunction, and blood-brain barrier disruption-play pivotal roles in mediating delayed brain injury and neurological deterioration. However, how these biological processes interact and contribute to heterogeneous outcomes remains poorly understood.

This multicenter study aims to elucidate the molecular mechanisms underlying post-rupture complications and prognosis in aSAH through integrative multi-omics and clinical data analysis. By combining genomic, transcriptomic, proteomic, metabolomic, and imaging-omic approaches using biospecimens such as blood, cerebrospinal fluid, urine, and other relevant tissues, this project seeks to identify key molecular pathways and biomarkers associated with secondary injury and outcome variation. The findings are expected to provide systematic insights into the biological basis of aSAH progression and establish a foundation for precision prediction and individualized management.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥18 years;
2. Confirmed diagnosis of aneurysmal subarachnoid hemorrhage (aSAH) by CTA, or DSA;
3. Aneurysm secured by either microsurgical clipping or endovascular coiling during hospitalization;
4. Time from onset to aneurysm treatment ≤ 72 hours;
5. Availability of biospecimens, including blood, cerebrospinal fluid (CSF), urine, or fecal samples collected during hospitalization;
6. Signed informed consent obtained from the patient or legal representative.

Exclusion Criteria:

1. History of previous intracranial aneurysm surgery or embolization;
2. Non-aneurysmal SAH, traumatic SAH, or perimesencephalic non-aneurysmal hemorrhage;
3. Presence of malignancy, severe hepatic or renal dysfunction, or other systemic diseases that may affect survival or biomarker expression;
4. Severe cardiorespiratory insufficiency or unstable medical condition precluding study participation;
5. Pregnancy or lactation;
6. Refusal to participate or withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult patients (≥18 years) with aneurysmal subarachnoid hemorrhage (aSAH) confirmed by CTA, or DSA, whose aneurysms are treated by microsurgical clipping or endovascular coiling within 72 hours after onset. Participants will be consecutively recruited from multiple tertiary neurosurgical centers.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) score for functional outcome | 3, 6, and 12 months after onset
  Functional outcome will be evaluated using the modified Rankin Scale (mRS), ranging from 0 (no symptoms) to 6 (death). Higher scores indicate greater disability. The distribution of mRS scores will be analyzed at predefined follow-up time points.

SECONDARY OUTCOMES:
Incidence of rebleeding | After onset, up to 30 days
  Rebleeding is defined as sudden clinical deterioration during postoperative hospitalization, accompanied by evidence of increased bleeding on serial CT scans.
Incidence of delayed cerebral ischemia (DCI) | After onset, up to 30 days
  DCI is defined as new focal neurological deficits or global neurological deterioration (a decrease of ≥2 points on the Glasgow Coma Scale) lasting more than 2 hours, after excluding intracranial hemorrhage, hydrocephalus, seizures, metabolic derangements, and infection, with or without radiological evidence of cerebral vasospasm.
Incidence of anemia | After onset, up to 30 days
  Anemia is defined as hemoglobin (HGB) < 120 g/L in adult males or < 110 g/L in adult females.Severity is categorized as: mild (HGB 90-120 g/L), moderate (60-90 g/L), severe (30-60 g/L), and very severe (<30 g/L).
Incidence of pneumonia | From enrollment to the end of follow-up at 3 months
  Pneumonia is defined as the presence of clinical indications such as fever, cough, purulent sputum, or positive chest radiographic findings consistent with pulmonary infection.
Incidence of deep vein thrombosis (DVT) | After onset, up to 30 days
  DVT is defined as thrombosis diagnosed by ultrasound or venography, with or without clinical symptoms such as limb pain or swelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided